CLINICAL TRIAL: NCT01981863
Title: Fibrinolysis Before Cardiopulmonary Bypass?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Fibrinolysis
Record Dates: First submitted 2013-09-19; First posted 2013-11-13 (Estimated); Results first posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-04

CONDITIONS: Pathologic Fibrinolysis
Keywords: cardiac surgery; cardiopulmonary bypass; fibrinolysis; thromboelastography; D-Dimers; antifibrinolytic agents
MeSH Terms: interventions — Aminocaproic Acid

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epsilonaminocaproic acid (Experimental): One arm: Epsilonaminocaproic acid 10 gr IV, followed by 1 gr/hr infusion Second arm: placebo
  Interventions: Drug: Epsilonaminocaproic acid
- Placebo, Antifibrinolytic activity (Placebo Comparator): Placebo: same IV volume as experimental arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Epsilonaminocaproic acid — One group receives Epsilonaminocaproic acid, 10 gr IV bolus, followed by 1 gr/hr. Second group receives placebo.
  Other Names: Amicar
  Arms: Epsilonaminocaproic acid
Drug: Placebo — Placebo administered in same volume as in experimental arm.
  Arms: Placebo, Antifibrinolytic activity

SUMMARY:
It is common practice to use antifibrinolytic agents before and during cardiopulmonary bypass. They are not without side effects. The investigators want to show that there is no proof of fibrinolysis in standard sternotomy cardiac surgery patients before cardiopulmonary bypass, and that antifibrinolytic agents should only be started on cardiopulmonary bypass.

DETAILED DESCRIPTION:
Double-blind, placebo controlled, prospective study in two groups of 20 patients. Control group (A) receives standard Epsilonaminocaproic acid treatment before cardiopulmonary bypass (10 gr loading dose, and 1 gr/hr infusion), and second group (B) receives placebo. Before start of Epsilonaminocaproic acid/placebo, D-Dimers and Thromboelastography are measured, repeated just before full heparinization. After heparinization group A receives placebo, and group B Epsilonaminocaproic acid.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, undergoing first time sternotomy for Coronary artery bypass grafting/Aortic valve replacement/aortic surgery

Exclusion Criteria:

* Resternotomy, renal insufficiency, deep hypothermia, age < 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter JA Van der Starre, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital & Clinics, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Epsilonaminocaproic Acid | Placebo, Antifibrinolytic Activity
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epsilonaminocaproic Acid | Placebo, Antifibrinolytic Activity | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (17) | 60 (15) | 58 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Di-Dimer Increase Before Cardiopulmonary Bypass
Description: Change in Di-dimer between preoperative value and value immediately before cardiopulmonary bypass in cardiac surgery patients.
Time Frame: 6 months
Population: D-Dimer from preoperative value and value immediately before cardiopulmonary bypass in cardiac surgery patients
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Epsilonaminocaproic Acid | Placebo, Antifibrinolytic Activity
Number analyzed (Participants) | 20 | 20
ng/mL
  Preoperative Value | 317 [200 to 2862] | 266 [200 to 1224]
  Immediately Before Cardiopulmonary Bypass | 317 [200 to 2689] | 291 [200 to 1206]
  Post cardiopulmonary bypass | 537 [200 to 3302] | 911 [266 to 3322]

2. Secondary Outcome: Value of Thromboelastography as Monitor of Fibrinolysis
Description: Thromboelastography may display if fibrinolysis is present
Time Frame: 6 months
Measure: Median (Full Range); unit: percentage of clot
Arm/Group | Epsilonaminocaproic Acid | Placebo, Antifibrinolytic Activity
Number analyzed (Participants) | 20 | 20
percentage of clot
  Preoperative Estimated Plasma Lysis | 0 [0 to 100] | 0 [0 to 100]
  Estimated Plasma Lysis Prior to Bypass | 0 [0 to 100] | 0 [0 to 100]
  Estimated Plasma Lysis Post Bypass | 0 [0 to 100] | 0 [0 to 100]

3. Other Pre Specified Outcome: Length of Time Between Incision and Cardiopulmonary Bypass
Description: Mean Length of Time from Incision to Cardiopulmonary Bypass
Time Frame: From incision to bypass, up to 3 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Epsilonaminocaproic Acid | Placebo, Antifibrinolytic Activity
Number analyzed (Participants) | 20 | 20
Minutes | 140 (63) | 165 (63)
Statistical Analysis 1: Comparison: Epsilonaminocaproic Acid vs Placebo, Antifibrinolytic Activity; Test type: Superiority or Other; p = 0.21, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Intraoperatively: From Induction to Post-Protamine administration, up to 12 hours
Groups:
- Epsilonaminocaproic Acid: One arm: Epsilonaminocaproic acid 10 gr IV, followed by 1 gr/hr infusion Second arm: placebo
  Epsilonaminocaproic acid: One group receives Epsilonaminocaproic acid, 10 gr IV bolus, followed by 1 gr/hr. Second group receives placebo.
  No adverse advents to report.
- Placebo, Antifibrinolytic Activity: Placebo: same IV volume as experimental arm
  Placebo: Placebo administered in same volume as in experimental arm.
  No adverse events to report.
Arm/Group | Epsilonaminocaproic Acid | Placebo, Antifibrinolytic Activity
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes